CLINICAL TRIAL: NCT00502515
Title: A Multi-center, Randomized, Double-blind, Placebo Controlled Study of the Effect of SSR180575 at Two Doses for 24 Weeks Treatment on the Rate of Regeneration of Epidermal Nerve Fibers in Patients With Mild Diabetic Peripheral Neuropathy
Brief Title: Dose-effect of SSR180575 in Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDY5807
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetes; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — SSR180575

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 25 mg SSR180575 (Experimental): orally once daily for 24 weeks
  Interventions: Drug: SSR180575
- 100 mg SSR180575 (Experimental): orally once daily for 24 weeks
  Interventions: Drug: SSR180575
- Placebo (Placebo Comparator): orally once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSR180575 — Oral, once daily dosing
  Arms: 100 mg SSR180575; 25 mg SSR180575
Drug: Placebo — Oral, once daily dosing
  Arms: Placebo

SUMMARY:
The primary objective of this sudy is to assess the effect of two doses of SSR180575 on the rate of regeneration of epidermal nerve fibers following denervation of the epidermal layer with capsaicin in patients with diabetes mellitus and mild peripheral neuropathy. Secondary objectives are to explore the efficacy of SSR180575 on clinical assessment, nerve function measures and to assess the tolerability and safety of SSR180575. The treatment period is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Diabetes Mellitus, type I or II, treated or untreated
* Diabetic neuropathy treated or untreated

Exclusion Criteria:

* Patients with unstable glycemic control
* Patients who have been hospitalized for a diabetes complication in the 3 months prior to randomization
* Patients with peripheral neuropathy attributable to any cause other than diabetes
* Non-measurable sural nerve sensory response on nerve conduction studies
* Amputation of any part of lower extremity
* Patients with a history of myocardial infarction or known coronary artery disease
* Grade III or IV heart failure on New York Heart Association criteria

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Rate of epidermal nerve fiber regeneration | 24 weeks

SECONDARY OUTCOMES:
Efficacy: change between baseline and 24 weeks of peripheral neuropathy assessed with nerve conduction studies, clinical evaluation, Total Neuropathy Score | 24 weeks
Safety: physical examination, clinical laboratories, adverse event reporting | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States